CLINICAL TRIAL: NCT01646398
Title: A Phase 3, Randomized, Modified Double-Blind, Active-Controlled Trial Evaluating The Safety, Tolerability, And Immunogenicity Of A 13-Valent Pneumococcal Conjugate Vaccine In Japanese Elderly Adults Aged 65 Years Old And Older Who Are Naive To Pneumococcal Vaccine
Brief Title: A Phase 3 Trial Evaluating the Safety, Tolerability, and Immunogenicity of a 13-valent Pneumococcal Conjugate Vaccine in Japanese Elderly Adults Aged 65 Years Old and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B1851088
Record Dates: First submitted 2012-05-10; First posted 2012-07-20 (Estimated); Results first posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-07

CONDITIONS: Pneumococcal Vaccines; Pneumococcal Conjugate Vaccine
Keywords: 13VPNC; 23VPS
MeSH Terms: interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- >= 65-year age group-13vPnC (Experimental)
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine
- >= 65-year age group-23vPS (Active Comparator)
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — A single dose (0.5 mL) will be administered intramuscularly into the deltoid muscle at visit 1.
  Other Names: 13vPnC
  Arms: >= 65-year age group-13vPnC
Biological: 23-valent pneumococcal polysaccharide vaccine — A single dose (0.5 mL) will be administered intramuscularly into the deltoid muscle at visit 1.
  Other Names: 23VPS
  Arms: >= 65-year age group-23vPS

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and immunogenicity of a single dose of 13-valent pneumococcal conjugate vaccine compared to a single dose of 23-valent pneumococcal polysaccharide vaccine in Japanese adults aged 65 years old and older.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Japanese male and female adults aged 65 years old and older at time of enrollment. Subjects with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease 12 weeks before receipt of the study vaccine, are eligible.
2. Male and female subjects of childbearing potential must agree to use a highly effective method of contraception throughout the study or for at least 28 days after the last dose of the study vaccine whichever is longer.

Exclusion Criteria:

1. History of severe adverse reaction including hypersensitivity such as anaphylaxis associated with a vaccine or vaccine component.
2. Previous vaccination with any licensed or experimental pneumococcal vaccine.
3. Documented Streptococcus pneumoniae infection within the past 5 years.
4. Residence in a nursing home, long-term care facility, or other institution or requirement of semiskilled nursing care.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 764 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Japan (8):
  - Medical Co.LTA PS Clinic, Fukuoka, Fukuoka
  - Seishinkai Inoue Hospital, Itoshima, Fukuoka
  - Yokohama Minoru Clinic, Yokohama, Kanagawa
  - Uzumasa Medical Clinic, Kyoto, Kyoto
  - Senbon Hospital, Osaka, Osaka
  - Oda Clinic, Shinjuku-ku, Tokyo
  - Sone Clinic, Shinjuku-ku, Tokyo
  - Medical Co. LTA Sumida Hospital, Sumida-ku, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1851088&StudyName=A%20Phase%203%20Trial%20Evaluating%20the%20Safety%2C%20Tolerability%2C%20and%20Immunogenicity%20of%20a%2013-valent%20Pneumococcal%20Conjugate%20Vaccine%20in%20Japanese%20Elde

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) administered as a 0.5 milliliter (mL) single dose intramuscularly on Day 1.
- 23vPS: 23-valent pneumococcal polysaccharide vaccine (23vPS) administered as a 0.5 mL single dose intramuscularly on Day 1.
Period: Overall Study
Arm/Group | 13vPnC | 23vPS
Started | 382 | 382
Completed | 381 | 382
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC | 23vPS | Total
Number analyzed (Participants) | 382 | 382 | 764
Age Continuous [Mean (Standard Deviation); unit: years] | 70.0 (4.08) | 69.7 (3.66) | 69.9 (3.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198 | 187 | 385
  Male | 184 | 195 | 379

OUTCOME MEASURES:

1. Primary Outcome: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for 12 Common Serotypes 1 Month After Vaccination
Description: Antibody-mediated serum OPA against each of the 12 pneumococcal serotypes (1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) was measured centrally using a quantitative functional microcolony OPA (mcOPA) assay. Results were expressed as OPA titers. OPA titers were logarithmically transformed for analysis; geometric means calculated and expressed as geometric mean titers (GMTs).
Time Frame: One month after vaccination
Population: Evaluable immunogenicity population:eligible participants, received study vaccine to which randomized, received no prohibited vaccines, had at least 1 valid and determinate assay result, had blood drawn within prescribed time frame and had no major protocol violations. n= number of participants with determinate OPA antibody titer to given serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC | 23vPS
Number analyzed (Participants) | 366 | 367
titer
  1 (n=366, 366) | 103 [84.6 to 125.5] | 78 [63.6 to 95.8]
  3 (n=365, 367) | 44 [38.1 to 51.5] | 61 [52.8 to 70.1]
  4 (n=360, 362) | 1016 [850.7 to 1213.2] | 392 [314.7 to 487.1]
  5 (n=350, 361) | 347 [282.3 to 425.6] | 118 [98.4 to 142.5]
  6B (n=360, 359) | 1995 [1689.3 to 2355.9] | 1440 [1223.5 to 1694.2]
  7F (n=365, 364) | 1901 [1642.8 to 2198.7] | 1361 [1153.3 to 1605.6]
  9V (n=365,358) | 858 [675.7 to 1089.5] | 379 [290.2 to 493.9]
  14 (n=363, 359) | 1028 [866.9 to 1217.9] | 1059 [896.6 to 1250.6]
  18C (n=366, 362) | 2015 [1675.4 to 2424.5] | 938 [752.7 to 1170.1]
  19A (n=365, 362) | 985 [841.5 to 1153.9] | 429 [358.0 to 513.2]
  19F (n=352, 357) | 773 [607.9 to 983.0] | 388 [305.6 to 491.8]
  23F (n=366, 363) | 456 [363.7 to 570.6] | 180 [143.1 to 226.1]
Statistical Analysis 1: Comparison: 13vPnC vs 23vPS; Serotype 1: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.3, 95% CI 2-sided [0.99 to 1.75]
Statistical Analysis 2: Comparison: 13vPnC vs 23vPS; Serotype 3: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 0.7, 95% CI 2-sided [0.59 to 0.89]
Statistical Analysis 3: Comparison: 13vPnC vs 23vPS; Serotype 4: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.6, 95% CI 2-sided [1.96 to 3.44]
Statistical Analysis 4: Comparison: 13vPnC vs 23vPS; Serotype 5: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.9, 95% CI 2-sided [2.22 to 3.86]
Statistical Analysis 5: Comparison: 13vPnC vs 23vPS; Serotype 6B: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.4, 95% CI 2-sided [1.10 to 1.75]
Statistical Analysis 6: Comparison: 13vPnC vs 23vPS; Serotype 7F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.4, 95% CI 2-sided [1.12 to 1.74]
Statistical Analysis 7: Comparison: 13vPnC vs 23vPS; Serotype 9V: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.3, 95% CI 2-sided [1.59 to 3.24]
Statistical Analysis 8: Comparison: 13vPnC vs 23vPS; Serotype 14: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 1.0, 95% CI 2-sided [0.77 to 1.23]
Statistical Analysis 9: Comparison: 13vPnC vs 23vPS; Serotype 18C: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.1, 95% CI 2-sided [1.61 to 2.86]
Statistical Analysis 10: Comparison: 13vPnC vs 23vPS; Serotype 19A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.3, 95% CI 2-sided [1.81 to 2.92]
Statistical Analysis 11: Comparison: 13vPnC vs 23vPS; Serotype 19F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.0, 95% CI 2-sided [1.42 to 2.79]
Statistical Analysis 12: Comparison: 13vPnC vs 23vPS; Serotype 23F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0.5; GMT Ratio = 2.5, 95% CI 2-sided [1.84 to 3.49]

2. Primary Outcome: Percentage of Participants Achieving At Least a 4-fold Rise in OPA Titers for Serotype 6A 1 Month After Vaccination
Description: For serotype 6A the percentage of participants achieving at least a 4-fold rise on the serotype-specific antibody titer from pre-vaccination to 1 month post-vaccination was computed along with exact, 2-sided 95% confidence interval for the proportion.
Time Frame: One month after vaccination
Population: Evaluable immunogenicity population. Here 'N' (number of participants analyzed) signifies participants with determinate fold rise of OPA antibody titer to serotype 6A.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 23vPS
Number analyzed (Participants) | 319 | 320
percentage of participants | 74.0 [68.8 to 78.7] | 47.2 [41.6 to 52.8]
Statistical Analysis 1: Comparison: 13vPnC vs 23vPS; Difference in proportions (13vPnC - 23vPS) expressed as a percentage presented along with exact, 2-sided 95%CI. Statistical significance was to be concluded if the lower bound of the 2-sided 95% CI was greater than 0; Test type: Superiority or Other; Difference in percentage = 26.8, 95% CI 2-sided [19.3 to 34.0]

3. Secondary Outcome: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for 12 Common Serotypes and Serotype 6A 1 Month After Vaccination
Description: Antibody-mediated serum OPA against each of the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) was measured centrally using a quantitative functional microcolonoy OPA (mcOPA) assay. Results were expressed as OPA titers. OPA titers were logarithmically transformed for analysis; geometric means calculated and expressed as geometric mean titers (GMTs).
Time Frame: One month after vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC | 23vPS
Number analyzed (Participants) | 366 | 367
titer
  1 (n=366, 366) | 103 [84.6 to 125.5] | 78 [63.6 to 95.8]
  3 (n=365, 367) | 44 [38.1 to 51.5] | 61 [52.8 to 70.1]
  4 (n=360, 362) | 1016 [850.7 to 1213.2] | 392 [314.7 to 487.1]
  5 (n=350, 361) | 347 [282.3 to 425.6] | 118 [98.4 to 142.5]
  6B (n=360, 359) | 1995 [1689.3 to 2355.9] | 1440 [1223.5 to 1694.2]
  7F (n=365, 364) | 1901 [1642.8 to 2198.7] | 1361 [1153.3 to 1605.6]
  9V (n=365,358) | 858 [675.7 to 1089.5] | 379 [290.2 to 493.9]
  14 (n=363, 359) | 1028 [866.9 to 1217.9] | 1059 [896.6 to 1250.6]
  18C (n=366, 362) | 2015 [1675.4 to 2424.5] | 938 [752.7 to 1170.1]
  19A (n=365, 362) | 985 [841.5 to 1153.9] | 429 [358.0 to 513.2]
  19F (n=352, 357) | 773 [607.9 to 983.0] | 388 [305.6 to 491.8]
  23F (n=366, 363) | 456 [363.7 to 570.6] | 180 [143.1 to 226.1]
  6A (n=360, 349) | 2122 [1790.9 to 2515.2] | 676 [542.4 to 841.7]
Statistical Analysis 1: Comparison: 13vPnC vs 23vPS; Serotype 1: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS). Statistical significance was to be concluded if the lower bound of the 2-sided 95% CI was greater than 1.0; Test type: Superiority or Other; GMT Ratio = 1.3, 95% CI 2-sided [0.99 to 1.75]
Statistical Analysis 2: Comparison: 13vPnC vs 23vPS; Serotype 3: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS). Statistical significance was to be concluded if the lower bound of the 2-sided 95% CI was greater than 1.0; Test type: Superiority or Other; GMT Ratio = 0.7, 95% CI 2-sided [0.59 to 0.89]
Statistical Analysis 3: Comparison: 13vPnC vs 23vPS; Serotype 4: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS). Statistical significance was to be concluded if the lower bound of the 2-sided 95% CI was greater than 1.0; Test type: Superiority or Other; GMT Ratio = 2.6, 95% CI 2-sided [1.96 to 3.44]
Statistical Analysis 4: Comparison: 13vPnC vs 23vPS; Serotype 5: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS). Statistical significance was to be concluded if the lower bound of the 2-sided 95% CI was greater than 1.0; Test type: Superiority or Other; GMT Ratio = 2.9, 95% CI 2-sided [2.22 to 3.86]
Statistical Analysis 5: Comparison: 13vPnC vs 23vPS; Serotype 6B: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS). Statistical significance was to be concluded if the lower bound of the 2-sided 95% CI was greater than 1.0; Test type: Superiority or Other; GMT Ratio = 1.4, 95% CI 2-sided [1.10 to 1.75]
Statistical Analysis 6: Comparison: 13vPnC vs 23vPS; Serotype 7F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS). Statistical significance was to be concluded if the lower bound of the 2-sided 95% CI was greater than 1.0; Test type: Superiority or Other; GMT Ratio = 1.4, 95% CI 2-sided [1.12 to 1.74]
Statistical Analysis 7: Comparison: 13vPnC vs 23vPS; Serotype 9V: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS). Statistical significance was to be concluded if the lower bound of the 2-sided 95% CI was greater than 1.0; Test type: Superiority or Other; GMT Ratio = 2.3, 95% CI 2-sided [1.59 to 3.24]
Statistical Analysis 8: Comparison: 13vPnC vs 23vPS; Serotype 14: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS). Statistical significance was to be concluded if the lower bound of the 2-sided 95% CI was greater than 1.0; Test type: Superiority or Other; GMT Ratio = 1.0, 95% CI 2-sided [0.77 to 1.23]
Statistical Analysis 9: Comparison: 13vPnC vs 23vPS; Serotype 18C: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS). Statistical significance was to be concluded if the lower bound of the 2-sided 95% CI was greater than 1.0; Test type: Superiority or Other; GMT Ratio = 2.1, 95% CI 2-sided [1.61 to 2.86]
Statistical Analysis 10: Comparison: 13vPnC vs 23vPS; Serotype 19A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS). Statistical significance was to be concluded if the lower bound of the 2-sided 95% CI was greater than 1.0; Test type: Superiority or Other; GMT Ratio = 2.3, 95% CI 2-sided [1.81 to 2.92]
Statistical Analysis 11: Comparison: 13vPnC vs 23vPS; Serotype 19F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS). Statistical significance was to be concluded if the lower bound of the 2-sided 95% CI was greater than 1.0; Test type: Superiority or Other; GMT Ratio = 2.0, 95% CI 2-sided [1.42 to 2.79]
Statistical Analysis 12: Comparison: 13vPnC vs 23vPS; Serotype 23F: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS). Statistical significance was to be concluded if the lower bound of the 2-sided 95% CI was greater than 1.0; Test type: Superiority or Other; GMT Ratio = 2.5, 95% CI 2-sided [1.84 to 3.49]
Statistical Analysis 13: Comparison: 13vPnC vs 23vPS; Serotype 6A: CI for the GMT ratio was calculated by the back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC - 23vPS). Statistical significance was to be concluded if the lower bound of the 2-sided 95% CI was greater than 2.0; Test type: Superiority or Other; GMT Ratio = 3.1, 95% CI 2-sided [2.38 to 4.14]

4. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination
Description: Local reactions reported using an electronic diary. Redness and swelling scaled as Any (redness present or swelling present); Mild (2.5 to 5.0 centimeters [cm]; Moderate (5.1 to 10.0 cm); Severe (>10 cm). Pain scaled as Any (pain present); Mild (awareness of pain; easily tolerated); Moderate (discomfort enough to cause interference with usual activity); Severe (incapacitating). Limitation of arm movement scaled as Any (limitation present); Mild (some limitation); Moderate (unable to move arm above head; able to move arm above shoulder); Severe (unable to move arm above shoulder).
Time Frame: Within 14 days after vaccination
Population: Safety population included all participants who received the study vaccine. 'N' (number of participants analyzed)=participants with known values for any local reaction. 'n'=number of participants with known values for specified local reaction for each group respectively. Participants may be represented in more than 1 category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 23vPS
Number analyzed (Participants) | 367 | 370
percentage of participants
  Redness: Any (n=355, 363) | 28.7 [24.1 to 33.7] | 10.5 [7.5 to 14.1]
  Redness: Mild (n=352, 362) | 22.2 [17.9 to 26.9] | 7.7 [5.2 to 11.0]
  Redness: Moderate (n=353, 360) | 17.3 [13.5 to 21.6] | 3.9 [2.1 to 6.4]
  Redness: Severe (n=349, 359) | 3.4 [1.8 to 5.9] | 0.3 [0.0 to 1.5]
  Swelling: Any (n=353, 360) | 21.5 [17.4 to 26.2] | 6.7 [4.3 to 9.8]
  Swelling: Mild (n=351, 360) | 16.5 [12.8 to 20.8] | 5.0 [3.0 to 7.8]
  Swelling: Moderate (n=351, 359) | 9.7 [6.8 to 13.3] | 2.5 [1.2 to 4.7]
  Swelling: Severe (n=349, 359) | 1.4 [0.5 to 3.3] | 0.3 [0.0 to 1.5]
  Pain: Any (n=362, 368) | 45.6 [40.4 to 50.9] | 38.3 [33.3 to 43.5]
  Pain: Mild (n=362, 368) | 45.3 [40.1 to 50.6] | 37.5 [32.5 to 42.7]
  Pain: Moderate (n=349, 361) | 2.9 [1.4 to 5.2] | 5.5 [3.4 to 8.4]
  Pain: Severe (n=348, 359) | 0.0 [0.0 to 1.1] | 1.4 [0.5 to 3.2]
  Limitation of arm movement: Any (n=355, 362) | 16.3 [12.6 to 20.6] | 16.9 [13.1 to 21.1]
  Limitation of arm movement: Mild (n=355, 361) | 15.5 [11.9 to 19.7] | 15.8 [12.2 to 20.0]
  Limitation of arm movement: Moderate(n=348, 360) | 1.1 [0.3 to 2.9] | 3.6 [1.9 to 6.1]
  Limitation of arm movement: Severe (n=348, 359) | 0.3 [0.0 to 1.6] | 1.7 [0.6 to 3.6]

5. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination
Description: Systemic events reported using an electronic diary. Systemic events are any fever greater than or equal to (>=) 37.5 degrees Celsius [C], fatigue, headache, chills, rash, vomiting, decreased appetite, new muscle pain, aggravated muscle pain, new joint pain, aggravated joint pain, use of medication to treat fever and use of medication to treat pain. All reports of fever >=39 degrees C in 13vPnC and 23vPS were confirmed as data entry errors.
Time Frame: Within 14 days after vaccination
Population: Safety population included all participants who received the study vaccine. 'N' (number of participants analyzed)=participants with known values for any systemic events. 'n'=number of participants with known values for specified systemic events for each group respectively. Participants may be represented in more than 1 category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 23vPS
Number analyzed (Participants) | 357 | 366
percentage of participants
  Fever >=37.5 to <38.5 degrees C (n=348, 359) | 2.6 [1.2 to 4.9] | 2.8 [1.3 to 5.1]
  Fever >=38.5 to <39 degrees C (n=348, 359) | 0.3 [0.0 to 1.6] | 0.3 [0.0 to 1.5]
  Fever >=39 to <=40 degrees C (n=348, 359) | 0.0 [0.0 to 1.1] | 0.6 [0.1 to 2.0]
  Fever >40 degrees C (n=348, 359) | 0.9 [0.2 to 2.5] | 0.0 [0.0 to 1.0]
  Fatigue (n=352, 362) | 17.3 [13.5 to 21.7] | 16.0 [12.4 to 20.2]
  Headache (n=351, 361) | 9.4 [6.6 to 12.9] | 11.6 [8.5 to 15.4]
  Chills (n=348, 359) | 2.9 [1.4 to 5.2] | 1.1 [0.3 to 2.8]
  Rash (n=350, 359) | 8.9 [6.1 to 12.3] | 3.6 [1.9 to 6.1]
  Vomiting (n=348, 359) | 1.1 [0.3 to 2.9] | 0.6 [0.1 to 2.0]
  Decreased appetite (n=348, 360) | 3.7 [2.0 to 6.3] | 5.0 [3.0 to 7.8]
  New muscle pain (n=354, 362) | 18.4 [14.5 to 22.8] | 17.4 [13.6 to 21.7]
  Aggravated muscle pain (n=350, 359) | 4.0 [2.2 to 6.6] | 3.9 [2.1 to 6.5]
  New joint pain (n=350, 359) | 7.7 [5.1 to 11.0] | 7.0 [4.6 to 10.1]
  Aggravated joint pain (n=349, 359) | 2.9 [1.4 to 5.2] | 3.1 [1.5 to 5.4]
  Use of medication to treat fever (n=348, 360) | 0.9 [0.2 to 2.5] | 2.2 [1.0 to 4.3]
  Use of medication to treat pain (n=348, 360) | 1.1 [0.3 to 2.9] | 2.8 [1.3 to 5.0]

ADVERSE EVENTS:
Time Frame: AEs/SAEs: recorded from signing of informed consent form to completion of study. Participants recorded pre-specified AEs in electronic diary:local reactions; systemic events; use of antipyretic medication (up to 14 days after vaccination).
Description: SAEs and AEs were grouped by system organ class and summarized. AEs included AEs collected in the electronic diary (local and systemic reactions; systematic assessment) and AEs collected on the case report form at each visit (nonsystematic assessment).
Arm/Group | 13vPnC | 23vPS
Serious Adverse Events (participants affected / at risk) | 1/382 | 0/382
Other Adverse Events (participants affected / at risk) | 211/382 | 166/382
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC (N=382) | 23vPS (N=382)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC (N=382) | 23vPS (N=382)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1
Injection site pain (General disorders) | 2 | 1
Injection site erythema (General disorders) | 2 | 0
Chills (General disorders) | 1 | 0
Feeling hot (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 0 | 1
Injection site pruritus (General disorders) | 1 | 0
Injection site swelling (General disorders) | 1 | 0
Vaccination site pruritus (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 8
Pharyngitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Redness (Any) (Skin and subcutaneous tissue disorders) | 102/355 | 38/363
Redness (Mild) (Skin and subcutaneous tissue disorders) | 78/352 | 28/362
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 61/353 | 14/360
Redness (Severe) (Skin and subcutaneous tissue disorders) | 12/349 | 1/359
Swelling (Any) (Skin and subcutaneous tissue disorders) | 76/353 | 24/360
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 58/351 | 18/360
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 34/351 | 9/359
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 5/349 | 1/359
Pain (Any) (Skin and subcutaneous tissue disorders) | 165/362 | 141/368
Pain (Mild) (Skin and subcutaneous tissue disorders) | 164/362 | 138/368
Pain (Moderate) (Skin and subcutaneous tissue disorders) | 10/349 | 20/361
Pain (Severe) (Skin and subcutaneous tissue disorders) | 0/348 | 5/359
Limitation of arm movement (Any) (Skin and subcutaneous tissue disorders) | 58/355 | 61/362
Limitation of arm movement (Mild) (Skin and subcutaneous tissue disorders) | 55/355 | 57/361
Limitation of arm movement (Moderate) (Skin and subcutaneous tissue disorders) | 4/348 | 13/360
Limitation of arm movement (Severe) (Skin and subcutaneous tissue disorders) | 1/348 | 6/359
Fever >=37.5 to <38.5 degrees C (General disorders) | 9/348 | 10/359
Fever >=38.5 to <39 degrees C (General disorders) | 1/348 | 1/359
Fever >=39 to <=40 degrees C (General disorders) | 0/348 | 2/359 — All reports of fever >=39 degrees C in 13vPnC and 23vPS were confirmed as data entry errors.
Fever >40 degrees C (General disorders) | 3/348 | 0/359 — All reports of fever >=39 degrees C in 13vPnC and 23vPS were confirmed as data entry errors.
Fatigue (General disorders) | 61/352 | 58/362
Headache (General disorders) | 33/351 | 42/361
Chills (General disorders) | 10/348 | 4/359
Rash (General disorders) | 31/350 | 13/359
Vomiting (General disorders) | 4/348 | 2/359
Decreased appetite (General disorders) | 13/348 | 18/360
New muscle pain (General disorders) | 65/354 | 63/362
Aggravated muscle pain (General disorders) | 14/350 | 14/359
New joint pain (General disorders) | 27/350 | 25/359
Aggravated joint pain (General disorders) | 10/349 | 11/359

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.